CLINICAL TRIAL: NCT03422640
Title: Open Label Trial Evaluating the Efficacy of Apremilast for the Treatment of Frontal Fibrosing Alopecia
Brief Title: Trial Evaluating the Efficacy of Apremilast for the Treatment of Frontal Fibrosing Alopecia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bellevue Dermatology (Other)
Collaborators: Celgene (Industry)
Responsible Party: Principal Investigator, Clive Liu, Director, Bellevue Dermatology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD1-1
Record Dates: First submitted 2018-01-23; First posted 2018-02-06 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Frontal Fibrosing Alopecia
Keywords: Frontal Fibrosing Alopecia; Apremilast
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Intervention Model Description: This is open label single side study involvement 20 patient treated with Apremilast. Each enrolled patient may be evaluated at by a dermatologist using the Lichen Planopilaris Activity Index and Frontal Fibrosing Alopecia Index. Other measures include physician global assessment, dermatology quality of life and patients analogue score for pruritus. Pt will have visits at Week 0,2,4,8,12,16,20,24
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm with apremilast (Experimental): Open label arm treating frontal fibrosing alopecia with apremilast
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Open label treatment with apremilast
  Other Names: Otezla

SUMMARY:
This is open label single side study involvement 20 patient treated with Apremilast. Each enrolled patient may be evaluated at by a dermatologist using the Lichen Planopilaris Activity Index and Frontal Fibrosing Alopecia Index. Other measures include physician global assessment, dermatology quality of life and patients analogue score for pruritus. Pt will have visits at Week 0,2,4,8,12,16,20,24

DETAILED DESCRIPTION:
Frontal fibrosing alopecia (FFA) is a chronic immune mediated inflammatory disease characterized by inflammation of the hair follicle and scaring hair loss. Clinically, FFA presents as a progressive recession of the hairline in a frontal temporal distribution. Evidence suggests that timely and effective management can prevent the permanent loss of hair. Unfortunately, most current treatment have been disappointing with poor efficacy or high risk profile. The available of a safe effective treatment for this disease remains an unmet need Apremilast is a novel phosphodiesterase 4 inhibitor currently FDA approved to treat psoriasis and is under investigation for other auto immune conditions. The medication has a good safety profile with no required laboratory monitoring. This study primarily aimsto determine whether Apremilast offers any benefit for this difficult to treatment population

ELIGIBILITY:
Inclusion Criteria:

1. Must be in general good health (except for disease under study) as judged by the Investigator, based on medical history, physical examination, clinical laboratories, and urinalysis. (NOTE: The definition of good health means a subject does not have uncontrolled significant co-morbid conditions).
2. Male or Female and is at least 18 years of age, at the time of enrollment.
3. Females of childbearing potential (FCBP)† must have a negative pregnancy test at Screening and Baseline. While on investigational product and for at least 28 days after taking the last dose of investigational product, FCBP who engage in activity in which conception is possible must use one of the approved contraceptive§ options described below: Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy; 3. OR Option 2: Male or female condom (latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]; PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide. Male subjects (including those who have had a vasectomy) who engage in activity in which conception is possible must use barrier contraception (male latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]) while on investigational product and for at least 28 days after the last dose of investigational product.

   * † A female of childbearing potential is a sexually mature female who 1) has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) consecutive months (that is, has had menses at any time during the preceding 24 consecutive months).
   * § The female subject's chosen form of contraception must be effective by the time the female subject is randomized into the study (for example, hormonal contraception should be initiated at least 28 days before randomization).
4. Patients with an established diagnosis of FFA based on the enrolling investigator's clinical judgment
5. Patients who have been treated and failed one standard therapy including

   * Topical steroids
   * Short course systemic steroids
   * Systemic antibiotics
6. Patients who are on stable dose of topical steroids or systemic antibiotics
7. Patient and/or legal guardian has voluntarily signed and dated an informed consent/patient authorization form approved by an Institutional Review Board (IRB)/Ethics Committee (EC) if applicable according to local law, after the nature of the study has been explained and the patient has had the opportunity to ask questions.

Exclusion Criteria:

1. Other than disease under study, any clinically significant (as determined by the Investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major disease that is currently uncontrolled.
2. Any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if he/she were to participate in the study.
3. Prior history of suicide attempt at any time in the subject's life time prior to screening or randomization, or major psychiatric illness requiring hospitalization within the last 3 years.
4. Pregnant or breast feeding.
5. Active substance abuse or a history of substance abuse within 6 months prior to Screening.
6. Malignancy or history of malignancy, except for: a. treated [ie, cured] basal cell or squamous cell in situ skin carcinomas; b. treated [ie, cured] cervical intraepithelial neoplasia (CIN) or carcinoma in situ of cervix with no evidence of recurrence within the previous 5 years.
7. Use of any investigational drug within 4 weeks prior to randomization, or 5 pharmacokinetic/pharmacodynamic half lives, if known (whichever is longer).
8. Prior treatment with apremilast.
9. Patient who have underlying chronic infections including HIV, Hep B and C.
10. History of uncontrolled depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-07-12 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Lichen Planopilaris index | Week 0 to 24, patient visit week0,2,4,8,12,16,20,24
  The weights given to the symptoms (30%), signs (30%), anagen pull test (25%), and presence of spreading (15%) led to the equation: LPPAI (0-10) = (pruritus + pain + burning)/3 + (scalp erythema + perifollicular erythema + perifollicular scale)/3 + 2.5 (pull test) + 1.5 (spreading/2).
  Symptoms and signs are recorded on a 4-point scale. The anagen pull test involves grasping a small group of 10 to 20 hairs between the thumb, second finger, and third finger at the scalp end of the hair shafts, and pulling away from the scalp with a slow, firm perpendicular force to slide the fingers to the ends of the hair. The result is recorded both as a binary value (0 for no anagen hairs and 1 for the presence of anagen hairs) and as anagen hairs/total hairs pulled. Last is the assessment of spreading, recorded as 0 (no spreading) versus 1 (indeterminate) versus 2 (spreading).
  Our primary endpoint is percentage change from baseline

SECONDARY OUTCOMES:
Physicians global assessment | Weeks 0 to 24, patient visit week 0,2,4,8,12,16,20,24
  Physicians global assessment This is a a five point scale used to measure the severity of the disease at the time of the physicians evaluation. 0-Clear, 1-Almost Clear, 2-Mild, 3-Moderate, 4-Severe The lower the score the better the score
Visual Analogue Scale Pruritus | Weeks 0 to 24, patient visit week 0,2,4,8,12,16,20,24
  Patient draws a line that best represent the severity of itch: this is continuous scale from 0-10, 0 being no itching and 10 being worst possible itching. Patient is to draw a line along the scale that represent the itch.
Frontal Fibrosing Alopecia Index | Weeks 0 to 24, patient visit weeks 0,2,4,8,12,16,20,24
  This is a scoring system recently proposed by Holmes et al from the British Nail and Hair society. FFASI was compiled in two forms: FFASI and FFASI B. FFASI utilizes clinical images of the entire hairline, divided into four sections. Alopecia severity is graded 1-5 based on hairline recession. In order that hairline recession comprises the greatest proportion of the assessment, each grade is weighted. Nonscalp hair loss (eyebrow, eyelash, limb and flexural) are scored, as are associated features (facial papules; cutaneous, nail and mucosal lichen planus;and generalized scalp lichen planopilaris). Scores for hairline recession, inflammatory band, nonscalp loss and associated features may be combined to give a maximum score of 100. FFASI B uses the same format, but rather than grading alopecia it permits user-defined measurement of each hairline section. We will look at mean change in FFASI compared to baseline
Dermatology Quality of Life (DLQI) (Appendix E) Dermatology Quality of Life (DLQI) (Appendix E) Dermatology Quality of Life (DLQI) | Weeks 0 to 24, patient visit weeks 0,2,4,8,12,16,20,24
  This is a questionnaire which measures how much a subjects skin problems affect his life over the last week. It is a series of 10 questions regarding various daily activities and each question consist of 4 responses from Very much, A lot, A little to Not at all. 0-being not at all or not relevant , 1-a little, 2-a lot, 3-very much in addition question 7, 3-prevent work or studying, the scores are added together for total score. Interpretation of score: 0-1 No affect on patient's life, 2-4 small affect on patient's life, 6-10 moderate affect on patient's life, 11-20 large on affect on patien's life, 21-30 extreme affect on patient's life

CONTACTS AND LOCATIONS:
Overall Officials: Clive Liu, MD, Study Director — Bellevue Dermatology
Locations (1):
- Bellevue Dermatology, Bellevue, Washington, United States

IPD SHARING:
Plan to Share IPD: No